CLINICAL TRIAL: NCT03209102
Title: Multimodal Study of the Emotional Regulation and Impulsivity Among Adolescents with Borderline Personality Disorder : Stress Reactivity and Functional Imaging
Brief Title: Emotional Regulation and Impulsivity Among Adolescents with Borderline Personality Disorder
Acronym: ADOLIMIS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C16-58
Record Dates: First submitted 2017-06-13; First posted 2017-07-06 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Borderline Personality Disorder; Adolescent Development
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPD adolescents (Experimental): Adolescents suffering from Borderline Personality Disorder. Clinical assessment, Stress Elicitation Experiment, Structural and Functional MRI, salivary collections of amylase and cortisol
  Interventions: Other: Clinical assessment; Behavioral: Stress elicitation experiment; Other: Structural and Functional MRI; Biological: salivary collections of amylase and cortisol
- Healthy controls adolescents (Experimental): Healthy controls adolescents. Clinical assessment, Stress Elicitation Experiment, Structural and Functional MRI, salivary collections of amylase and cortisol
  Interventions: Other: Clinical assessment; Behavioral: Stress elicitation experiment; Other: Structural and Functional MRI; Biological: salivary collections of amylase and cortisol

INTERVENTIONS:
Other: Clinical assessment — * Self-assessments based on questionnaires : Strengths and Difficulties Questionnaire - Development and Well-Being Assessment (SDQ-DAWBA) ; Pubertal Development Scale ; Life Events Questionnaire ; Childhood Trauma Questionnaire ; Abbreviated - Diagnostic Instrument for Borderline (Ab-DIB) ; Beck Depression Inventory ; Socio-demographic questionnaire)
  * and clinical evaluation by a psychiatrist : Mini-International Neuropsychiatric Interview (MINI); Global Assessment of Functioning
Behavioral: Stress elicitation experiment — The stress elicitation experiment is based on a time-constrained mental arithmetic test in the presence of an observer. The task usually lasts about 30 minutes.
  During the task, the investigators will monitor: neuro-vegetative parameters (skin conductance, temperature, respiratory and cardiac frequencies, and VNA) ; biological parameters : salivary Cortisol and Amylase before test (baseline), 15 min and 30 min after testing (respectively corresponding to Reactivity and Recovery) ; micro-behavioral cues extracted from 2D video and 3D sensors (Microsoft Kinect).
Other: Structural and Functional MRI — Structural and Functional Magnetic Resonance Imaging (MRI). The functional acquisition will last 20 minutes and the structural acquisition 18 minutes. All MR image acquisition methodologies are already functioning on the 3 Tesla Prisma machine within the ICM(Brain and Spine Institute), Salpetriere. The fMRI session will provide three types of data: (1) task-related activity to probe the striato-limbic and prefrontal regions, (2) resting state connectivity to examine the integrity of canonical networks, and (3) MR structural images to measure regional volumes of key functional nodes.
  For the task-related fMRI study, the investigators will use the monetary incentive delay task that reliably elicit an activation in known functional networks underlying reward anticipation/outcome.
Biological: salivary collections of amylase and cortisol — Collection of saliva samples of cortisol and amylase repeated three times

SUMMARY:
This study aims to better understand the behavioral, neurobiological and hormonal underpinnings of stress and reward reactivity of adolescents suffering from borderline personality disorder compared to healthy adolescents by a multimodal approach based on clinical assessments, structural and functional mri and experimental acute stress exposure.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a severe condition associated with intense emotional and behavioral responses to stressful events, impulsivity, and risk-taking behavior. It has been shown to begin in adolescence. However, very few studies have addressed the physiopathology of BPD in adolescents. In order to gather rational information for targeted care, the heterogeneity of BPD determinants needs to be disentangled. To this aim, a multimodal approach to BPD dimensional aspects is proposed.

BPD adolescents will be compared to typically developing controls in two complementary experimental designs: (1) Monitoring of neurovegetative, hormonal and body motion responses to an acute stress, with the hypothesis that stress reactivity might account for the physiopathology of the disorder; (2) Structural and functional imaging (fMRI BOLD) in the context of a reward processing task to delineate the neural/functional basis of BPD risk taking behavior.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent subject: 13 years ≤ age ≤ 18years
* Affiliation to social welfare
* Informed consent to participate in the protocol, consent signed by the major subject or by one of the legal guardians if the subject is a minor
* Diagnosis of borderline personality disorder according to Diagnostic and Statistical Manual of Mental Disorders 5 (DSM-5) and Abbreviated- Diagnostic Interview of Borderline Personality Disorder (Ab-DIB)
* Somatic and intellectual state compatible with blood sampling and MRI examination

Exclusion Criteria:

* Non-affiliation to social welfare
* Refusal to give consent and / or to sign informed consent by the subject or his or her legal guardian if the subject is a minor
* Somatic pathology in progress, or pregnancy (urine test of pregnancy in case of doubt)
* Contraindication to magnetic resonance imaging:
* Presence of a ferromagnetic foreign body
* Subject carrying a pacemaker
* Subject carrying ventricular bypass valves
* Claustrophobic topic
* Subject suffering from the following diseases:
* Intellectual impairment Intellectual Quotient (IQ) <70,
* Claustrophobia,
* Obsessive Compulsive Disorder,
* Tic Disorder,
* Autism Spectrum Disorder,
* Attention Deficit Disorder with or without Hyperactivity,
* Bipolar disorder,
* Schizophrenia

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 66 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2026-01-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between subjective and objective acute stress experience in BPD Adolescents vs Healthy controls | up to 3 months
  Comparing subjective (by self-assessment) and objective response to acute stress by measuring the biological (stress hormones and enzymes) and neurovegetative responses to stress and assessing the motor responses to stress by using novel approaches based on specific machine learning algorithms.
Investigating the neural correlates and modulation of motivation and impulsivity using structural and task-based fMRI | up to 3 months
  The fMRI session will provide three types of data: (1) task-related activity to probe the striato-limbic and prefrontal regions, (2) resting state connectivity to examine the integrity of canonical networks, and (3) MR structural images to measure regional volumes of key functional nodes. For the task-related fMRI study, the investigators will use the monetary incentive delay task that reliably elicit an activation in known functional networks underlying reward anticipation/outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Pôle recherche clinique, Paris, France

IPD SHARING:
Plan to Share IPD: No